CLINICAL TRIAL: NCT00307606
Title: Does a Single Steroid Injection Reduce the Formation of Postmastectomy Seroma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: seromprotocol
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2007-09-06 (Estimated); Status verified 2005-12

CONDITIONS: Breast Neoplasms; Mastectomy
Keywords: Mastectomy; Seroma; Breast cancer; Glucocorticoid
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Solu-medrol 125 mg

SUMMARY:
Background Seroma formation is a common problem after mastectomy. The incidence various between 30% to 92%. It is often an ongoing problem after removal of the suction drain, and repeated skin puncture is necessary to remove the seroma. In addition to many ambulatory visits this also leads to an increased risk of infection, and the adjuvant treatment can be delayed for several weeks

Different procedures have been tried to avoid seroma formation. Among these are for ex. : immobilisation of the arm and shoulder after mastectomy, different drain regimens, closing of the dead space of the cavity, different chemical substances as thrombin, tranexamacid and fibrin. Non of these results has been successful.

Seroma formation is most likely the result of the inflammatory response due to wound healing. In the seroma fluid several factors have been detected that support this assumption. These factors are: high levels of IgG, leucocytes, granulocytes, proteinases, proteinases inhibitors, different kinds of cytokines ( tPA, uPA,, uPAR, PAI-1, PAI-2, IL-6 og IL-1).

On the basis of this, an inhibition of the inflammatory response might result in a decrease of seroma formation, and perhaps improve quality of life after mastectomy.

Steroids inhibit the inflammatory response for example by inhibition of the cytokine function. It has been shown that a high single dose of steroid infusion (30mg/kg solu-medrol) inhibits the normal IL 6 response after colon resection. Newer studies have shown that even at a lower dose the inflammatory response is inhibited. In several studies of head and neck surgery the oedema in surgical area is reduced after a single dose of 125 mg solumedrol. It is precisely this effect of reduced fluid formation we want to obtain in our study. We have therefore chosen to use a single dose of 125 mg of solumedrol in this study. Even at the largest single dose of glucocorticoids there have not been seen any increasing in surgical complications.

The aim of the study: To find out whether single dose of glucocorticoid can reduce the seroma formation after mastectomy

Study design : A randomised pilot study, with 2 x 20 patients. 125 mg solumedrol is given 1,5 hours before surgery in 20 patients, and the other 20 patients are the control group

Inclusion criteria: Women with primary breast cancer, undergoing a mastectomy with either sentinel node biopsy or complete axillary dissection.

DETAILED DESCRIPTION:
Background Seroma formation is a common problem after mastectomy. The incidence various between 30% to 92%. It is often an ongoing problem after removal of the suction drain, and repeated skin puncture is necessary to remove the seroma. In addition to many ambulatory visits this also leads to an increased risk of infection, and the adjuvant treatment can be delayed for several weeks

Different procedures have been tried to avoid seroma formation. Among these are for ex. : immobilisation of the arm and shoulder after mastectomy, different drain regimens, closing of the dead space of the cavity, different chemical substances as thrombin, tranexamacid and fibrin. Non of these results has been successful.

Seroma formation is most likely the result of the inflammatory response due to wound healing. In the seroma fluid several factors have been detected that support this assumption. These factors are: high levels of IgG, leucocytes, granulocytes, proteinases, proteinases inhibitors, different kinds of cytokines ( tPA, uPA,, uPAR, PAI-1, PAI-2, IL-6 og IL-1).

On the basis of this, an inhibition of the inflammatory response might result in a decrease of seroma formation, and perhaps improve quality of life after mastectomy.

Steroids inhibit the inflammatory response for example by inhibition of the cytokine function. It has been shown that a high single dose of steroid infusion (30mg/kg solu-medrol) inhibits the normal IL 6 response after colon resection. Newer studies have shown that even at a lower dose the inflammatory response is inhibited. In several studies of head and neck surgery the oedema in surgical area is reduced after a single dose of 125 mg solumedrol. It is precisely this effect of reduced fluid formation we want to obtain in our study. We have therefore chosen to use a single dose of 125 mg of solumedrol in this study. Even at the largest single dose of glucocorticoids there have not been seen any increasing in surgical complications.

The aim of the study: To find out whether single dose of glucocorticoid can reduce the seroma formation after mastectomy

Study design : A randomised pilot study, with 2 x 20 patients. 125 mg solumedrol is given 1,5 hours before surgery in 20 patients, and the other 20 patients are the control group

Inclusion criteria: Women with primary breast cancer, undergoing a mastectomy with either sentinel node biopsy or complete axillary dissection.

ELIGIBILITY:
Inclusion Criteria:

* Women with primary breast cancer, planned for a mastectomy with and axillary dissection.
* Age over 18 years
* signed informed consent.

Exclusion Criteria:

* Men
* Treatment with glucocorticoids within the last month before surgery, including inhalation products
* Pregnant.
* Not able to speak danish
* Severe heart disease
* Treatment with carbamazepine, phenytoin, phenobarbital, rifampicin, salicylates and ciclosporin
* Uræmia
* Diabetes
* Other medical conditions, evaluated by the investigator, that make tke patient unfit for participation
* previous psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-12; Study Completion 2007-12

PRIMARY OUTCOMES:
seroma formation

CONTACTS AND LOCATIONS:
Overall Officials: Christen Axelsson, Principal Investigator
Locations (1):
- Herlev Hospital, breast surgery, Herlev, Copenhagen, Denmark

REFERENCES:
- [Background] Burak WE Jr, Goodman PS, Young DC, Farrar WB. Seroma formation following axillary dissection for breast cancer: risk factors and lack of influence of bovine thrombin. J Surg Oncol. 1997 Jan;64(1):27-31. doi: 10.1002/(sici)1096-9098(199701)64:13.0.co;2-r. PMID 9040797
- [Background] Watt-Boolsen S, Jacobsen K, Blichert-Toft M. Total mastectomy with special reference to surgical technique, extent of axillary dissection and complications. Acta Oncol. 1988;27(6A):663-5. doi: 10.3109/02841868809091765. PMID 3219219
- [Background] Jeffrey SS, Goodson WH 3rd, Ikeda DM, Birdwell RL, Bogetz MS. Axillary lymphadenectomy for breast cancer without axillary drainage. Arch Surg. 1995 Aug;130(8):909-12; discussion 912-3. doi: 10.1001/archsurg.1995.01430080111018. PMID 7632155
- [Background] Kumar S, Lal B, Misra MC. Post-mastectomy seroma: a new look into the aetiology of an old problem. J R Coll Surg Edinb. 1995 Oct;40(5):292-4. PMID 8523301
- [Background] Porter KA, O'Connor S, Rimm E, Lopez M. Electrocautery as a factor in seroma formation following mastectomy. Am J Surg. 1998 Jul;176(1):8-11. doi: 10.1016/s0002-9610(98)00093-2. PMID 9683123
- [Background] Schultz I, Barholm M, Grondal S. Delayed shoulder exercises in reducing seroma frequency after modified radical mastectomy: a prospective randomized study. Ann Surg Oncol. 1997 Jun;4(4):293-7. doi: 10.1007/BF02303577. PMID 9181227
- [Background] Browse DJ, Goble D, Jones PA. Axillary node clearance: who wants to immobilize the shoulder? Eur J Surg Oncol. 1996 Dec;22(6):569-70. doi: 10.1016/s0748-7983(96)92164-2. PMID 9005140
- [Background] Barwell J, Campbell L, Watkins RM, Teasdale C. How long should suction drains stay in after breast surgery with axillary dissection? Ann R Coll Surg Engl. 1997 Nov;79(6):435-7. PMID 9422871
- [Background] Liu CD, McFadden DW. Overnight closed suction drainage after axillary lymphadenectomy for breast cancer. Am Surg. 1997 Oct;63(10):868-70. PMID 9322660
- [Background] Bonnema J, van Geel AN, Ligtenstein DA, Schmitz PI, Wiggers T. A prospective randomized trial of high versus low vacuum drainage after axillary dissection for breast cancer. Am J Surg. 1997 Feb;173(2):76-9. doi: 10.1016/S0002-9610(96)00416-3. PMID 9074367
- [Background] Medwid A. A new and quick method for treating postmastectomy seromas. Surg Gynecol Obstet. 1992 Feb;174(2):161-2. PMID 1734578
- [Background] Tadych K, Donegan WL. Postmastectomy seromas and wound drainage. Surg Gynecol Obstet. 1987 Dec;165(6):483-7. PMID 3686312
- [Background] Holcombe C, West N, Mansel RE, Horgan K. The satisfaction and savings of early discharge with drain in situ following axillary lymphadenectomy in the treatment of breast cancer. Eur J Surg Oncol. 1995 Dec;21(6):604-6. doi: 10.1016/s0748-7983(95)95133-4. PMID 8631403
- [Background] Coveney EC, O'Dwyer PJ, Geraghty JG, O'Higgins NJ. Effect of closing dead space on seroma formation after mastectomy--a prospective randomized clinical trial. Eur J Surg Oncol. 1993 Apr;19(2):143-6. PMID 8491318
- [Background] O'Dwyer PJ, O'Higgins NJ, James AG. Effect of closing dead space on incidence of seroma after mastectomy. Surg Gynecol Obstet. 1991 Jan;172(1):55-6. PMID 1985342
- [Background] Chilson TR, Chan FD, Lonser RR, Wu TM, Aitken DR. Seroma prevention after modified radical mastectomy. Am Surg. 1992 Dec;58(12):750-4. PMID 1456600
- [Background] Oertli D, Laffer U, Haberthuer F, Kreuter U, Harder F. Perioperative and postoperative tranexamic acid reduces the local wound complication rate after surgery for breast cancer. Br J Surg. 1994 Jun;81(6):856-9. doi: 10.1002/bjs.1800810621. PMID 8044602
- [Background] Uden P, Aspegren K, Balldin G, Garne JP, Larsson SA. Fibrin adhesive in radical mastectomy. Eur J Surg. 1993 May;159(5):263-5. PMID 8103359
- [Background] Wang JY, Goodman NC, Amiss LR Jr, Nguyen DH, Rodeheaver GT, Moore MM, Morgan RF, Abbott RD, Spotnitz WD. Seroma prevention in a rat mastectomy model: use of a light-activated fibrin sealant. Ann Plast Surg. 1996 Oct;37(4):400-5. doi: 10.1097/00000637-199610000-00009. PMID 8905048
- [Background] Harada RN, Pressler VM, McNamara JJ. Fibrin glue reduces seroma formation in the rat after mastectomy. Surg Gynecol Obstet. 1992 Nov;175(5):450-4. PMID 1440175
- [Background] Watt-Boolsen S, Nielsen VB, Jensen J, Bak S. Postmastectomy seroma. A study of the nature and origin of seroma after mastectomy. Dan Med Bull. 1989 Oct;36(5):487-9. PMID 2509147
- [Background] Baker EA, Leaper DJ. Proteinases, their inhibitors, and cytokine profiles in acute wound fluid. Wound Repair Regen. 2000 Sep-Oct;8(5):392-8. doi: 10.1111/j.1524-475x.2000.00392.x. PMID 11115151
- [Background] Doolin EJ, Tsuno K, Strande LF, Santos MC. Pharmacologic inhibition of collagen in an experimental model of subglottic stenosis. Ann Otol Rhinol Laryngol. 1998 Apr;107(4):275-9. doi: 10.1177/000348949810700402. PMID 9557759
- [Background] Schulze S, Andersen J, Overgaard H, Norgard P, Nielsen HJ, Aasen A, Gottrup F, Kehlet H. Effect of prednisolone on the systemic response and wound healing after colonic surgery. Arch Surg. 1997 Feb;132(2):129-35. doi: 10.1001/archsurg.1997.01430260027005. PMID 9041914
- [Background] Holte K, Kehlet H. Perioperative single-dose glucocorticoid administration: pathophysiologic effects and clinical implications. J Am Coll Surg. 2002 Nov;195(5):694-712. doi: 10.1016/s1072-7515(02)01491-6. No abstract available. PMID 12437261
- [Background] Sauerland S, Nagelschmidt M, Mallmann P, Neugebauer EA. Risks and benefits of preoperative high dose methylprednisolone in surgical patients: a systematic review. Drug Saf. 2000 Nov;23(5):449-61. doi: 10.2165/00002018-200023050-00007. PMID 11085349
- [Background] Apte RN, Voronov E. Interleukin-1--a major pleiotropic cytokine in tumor-host interactions. Semin Cancer Biol. 2002 Aug;12(4):277-90. doi: 10.1016/s1044-579x(02)00014-7. PMID 12147202
- [Background] Mettler L, Salmassi A, Heyer M, Schmutzier A, Schollmeyer T, Jonat W. Perioperative levels of interleukin-1beta and interleukin-6 in women with breast cancer. Clin Exp Obstet Gynecol. 2004;31(1):20-2. PMID 14998180
- [Background] Khan AL, Larsen F, Heys SD, Eremin O. Peri-operative acute phase response and cytokine releasein women with breast cancer: modulation bypolyadenylic-polyuridylic acid. Eur J Surg Oncol. 1999 Dec;25(6):574-9. doi: 10.1053/ejso.1999.0709. PMID 10556002
- [Background] Yokoe T, Iino Y, Morishita Y. Trends of IL-6 and IL-8 levels in patients with recurrent breast cancer: preliminary report. Breast Cancer. 2000;7(3):187-90. doi: 10.1007/BF02967458. PMID 11029796
- [Background] DeMichele A, Martin AM, Mick R, Gor P, Wray L, Klein-Cabral M, Athanasiadis G, Colligan T, Stadtmauer E, Weber B. Interleukin-6 -174G-->C polymorphism is associated with improved outcome in high-risk breast cancer. Cancer Res. 2003 Nov 15;63(22):8051-6. PMID 14633738
- [Background] Nishimura R, Nagao K, Miyayama H, Matsuda M, Baba K, Matsuoka Y, Yamashita H, Fukuda M, Mizumoto T, Hamamoto R. An analysis of serum interleukin-6 levels to predict benefits of medroxyprogesterone acetate in advanced or recurrent breast cancer. Oncology. 2000 Aug;59(2):166-73. doi: 10.1159/000012155. PMID 10971177
- [Background] Stewart T, Tsai SC, Grayson H, Henderson R, Opelz G. Incidence of de-novo breast cancer in women chronically immunosuppressed after organ transplantation. Lancet. 1995 Sep 23;346(8978):796-8. doi: 10.1016/s0140-6736(95)91618-0. PMID 7674744
- [Background] Guth AA. Breast cancer and human immunodeficiency virus infection: issues for the 21st century. J Womens Health (Larchmt). 2003 Apr;12(3):227-32. doi: 10.1089/154099903321667564. PMID 12804353